CLINICAL TRIAL: NCT00534521
Title: Posterior Tibial Nerve Stimulation vs. Sham
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2007-145
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; posterior tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment Arm (Active Comparator): Subjects will have their leg and foot draped to remain blinded to the test. They will be in a supine position with the knees abducted and flexed. The medial aspect of the lower extremity is palpated and a needle insertion site is identified. Between the posterior margin of the tibia and the soleus muscle, an acupuncture-like needle is inserted. An adhesive grounding pad is placed on the bottom of the foot just below the smallest toe. The needle and grounding pad are connected to the stimulator and the stimulation is increased as tolerated.
  Interventions: Device: Posterior Tibial Nerve Device
- Sham Arm (Sham Comparator): Since subjects with the PTNS will feel foot stimulation, the sham was devised to mimic this feeling without the tibial nerve being stimulated. Again the leg and foot will be draped and out of view from the subject. The medial aspect of the lower extremity is palpated (Figure 4) and the tibial nerve site is identified approximately 5 cm cephalad from the medial malleolus. A Streitberger needle is used at the tibial nerve insertion site to simulate needle placement without puncturing the skin. The needle will be taped in place as in the PTNS procedure. The "grounding pad" will be a gel electrode pad from a TENS unit device that is placed on the bottom of the foot just below the smallest toe.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Posterior Tibial Nerve Device — The PTNS device (Urgent® PC) is a minimally invasive neuromodulation system designed to deliver retrograde access to the sacral nerve through percutaneous electrical stimulation of the tibial nerve (PTNS). It is a combination of a stimulator and a lead set. The stimulator is a battery powered, external pulse generator and is designed, constructed, and manufactured for multiple use in conjunction with the lead set. The lead set (comprised of the lead wires, needle electrode, and alcohol pad) transfers the electrical current from the stimulator to the tibial nerve via the needle electrode. The tibial nerve travels up the leg to the sacral nerve plexus which regulates the bladder and pelvic floor function.
  Other Names: PTNS device; Urgent® PC
  Arms: Active Treatment Arm
Device: Sham — This 2- piece needle, comprised of a needle handle and blunt-tip shaft feels like a slight prick when touched to the skin. However the shaft retracts as it appears to enter the skin but the skin is not punctured. The Streitberger needle specifically activates the dorsolateral prefrontal cortex, which is associated with the placebo effect.
  Other Names: Streitberger needle
  Arms: Sham Arm

SUMMARY:
The overall goal of this research is to determine the efficacy of a sham for posterior tibial nerve stimulation (PTNS). This novel design is needed in order to have a sham treatment that is similar to the actual treatment. The PTNS is used to treat urgency and frequency in people with overactive bladder (OAB). Until research is done using a sham component, we are unable to ascertain if the current use of PTNS is due to a placebo effect.

DETAILED DESCRIPTION:
Subjects will be healthy volunteers who are recruited by word of mouth. At their office visit with the Nurse Practitioner (NP), the subject's history and medication list will be reviewed.

The NP will randomize subjects into groups: one group with the PTNS on the right and sham on the left; the other group with the PTNS on the left and sham on the right. There will be a maximum of 30 subjects tested, and up to 50 people screened. The subjects will have 1 session for the testing of the PTNS vs sham that will include 15 minutes of stimulation as noted below. All participants will be blinded to the therapy they receive as described below.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects >18 years of age
* Female subjects will be menopausal, or have had a tubal ligation or hysterectomy.
* Capable of giving informed consent
* Capable and willing to follow study related procedures

Exclusion Criteria:

* Pregnancy
* InterStim
* Bion
* TENS
* The subject is deemed unsuitable for enrollment in this study by the investigators based on their history or physical examination (including bleeding disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to determine the efficacy of a sham for posterior tibial nerve stimulation (PTNS). | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States